CLINICAL TRIAL: NCT02419638
Title: Comparison of Rebif Compared to Tecifdera on Six-month Outcomes in Patients With Relapsing-remitting MS
Status: Withdrawn | Type: Observational
Why Stopped: Collaborative decision between study PI and sponsor.
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: EMD Serono (Industry)
Responsible Party: Principal Investigator, Tanuja Chitnis, Attending Neurologist, Assoc. Professor of Neurology, Brigham and Women's Hospital
Other Study IDs: 2015P000242
Record Dates: First submitted 2015-04-14; First posted 2015-04-17 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-02

CONDITIONS: Multiple Sclerosis
Keywords: relapsing-remitting MS; lesions; treatment
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interferon beta-1a; Dimethyl Fumarate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Randomized Treatment Arm: Rebif: 120 patients treated with Rebif (IFN β-1a subcutaneous three times per week)
  Interventions: Drug: Rebif (IFN β-1a subcutaneous three times per week)
- Randomized Treatment Arm: Tecfidera: 120 patients treated with Tecfidera (dimethyl fumarate)
  Interventions: Drug: Tecifdera (dimethyl fumarate)

INTERVENTIONS:
Drug: Rebif (IFN β-1a subcutaneous three times per week)
  Groups: Randomized Treatment Arm: Rebif
Drug: Tecifdera (dimethyl fumarate)
  Groups: Randomized Treatment Arm: Tecfidera

SUMMARY:
To compare two commonly used MS medications, IFN β-1a subcutaneous three times per week (Rebif) and oral twice daily dimethyl fumarate (Tecfidera), on mean number of new or enlarging T2 lesions at 6 months in adults with relapsing-remitting multiple sclerosis who are prescribed these medications and receive a 6 month MRI scan as standard of care.

DETAILED DESCRIPTION:
Primary objective To compare two commonly used MS medications, IFN β-1a subcutaneous three times per week (Rebif) and oral twice daily dimethyl fumarate (Tecfidera), on mean number of new or enlarging T2 lesions at 6 months in adults with relapsing-remitting multiple sclerosis who are prescribed these medications and receive a 6 month MRI scan as standard of care.

Key secondary objective To compare Rebif vs. Tecfidera in reducing the T2 lesion volume, number of T1 black holes, gadolinium-enhancing lesions, brain parenchymal fraction, brain white matter fraction and brain gray matter fraction on the 6 month MRI.

Other secondary objectives

* To compare the two treatments on the following clinical efficacy measures which are routinely obtained as part of our clinical practice: Expanded disability status score (EDSS), ambulation index (AI), disease steps and number of relapses. In addition we will obtain the MSFC-4, which in addition to the AI which is routinely done, will include the symbol digit modalities test (SDMT), low contrast visual acuity, and 9 hole peg test.
* To compare adherence to the two treatments using an adherence question.

Tertiary objectives

* To compare the two treatments on optical coherence tomography (OCT) and visual acuity measures.
* To compare the following patient reported outcomes: MSQOL-54 (MSQOL54), Modified MOS Social Support Survey (MSSS), Modified Fatigue Impact Scale (MFIS), Center for Epidemiological Studies Depression Scale (CES-D).
* To compare cognitive function using the brief repeatable battery of neuropsychological tests in Multiple Sclerosis (BRB) which includes the following cognitive measures: Symbol Digit Modalities Test (SDMT), Selective Reminding Test (SRT), 10/36 Spatial Recall Test (10/36), Controlled Oral Word Association Test (COWAT).
* To compare the following Pharmacoeconomic outcomes: Healthcare Utilization and Costs, QUALY, Unscheduled visits (office, ER, hospital), out-of-pocket expenses (e.g., durable medical equipment, copays), Work Productivity and Activity Impairment (WPAI), Treatment satisfaction questionnaire (Treatment Satisfaction for Medication Questionnaire (TSQM))

Design: The study is a single center, 6-month, randomized, parallel-group, single blind study to compare two FDA approved treatments for MS (Rebif and Tecfidera) in adults with relapsing-remitting MS. 120 subjects will be treated with each medication (total 240 patients). Randomization will ensure balanced patient groups and prevent bias. Patients will be prescribed the medication by their treating physician who will follow the patient in a open fashion as part of standard of care for MS including obtaining MRI imaging at 6 months. At 6 months, patients will have a neurologic exam by an independent examining physician and administration of questionaires by study staff blinded to their treatment.

Methods: Relapsing-remitting patients beginning medication and deemed suitable for treatment with Rebif or Tecfidera as part of standard of care for MS will be explained the nature of the study, after which informed consent will be obtained. They will undergo a baseline visit and then randomized to one of the two treatments. Blood samples for biomarker studies will be collected at the baseline visit and at 6 months. MRI is obtained prior to therapy and at 6 months as part of standard of care. Following the completion of the 6 month study period, subjects are able to continue on either of the two treatments or switch to another agent according to their own preference and following discussions with their treating MS neurologist.

Subjects who discontinue treatments prior to the 6 month period are free to begin another therapy. Upon discontinuation of treatment, subjects will complete the end of study (EOS) visit as soon as possible and will be followed for the duration of the 6-month treatment phase.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects aged 18-65 years old, inclusive.
2. A diagnosis of MS as defined by the McDonald 2010 criteria for MS.
3. Relapsing form of MS, defined as at least one relapse in the prior 5 years.
4. Expanded Disability Status Scale (EDSS) score of 0 to 5.5, inclusive.
5. English language skills adequate for the completion of questionnaires and cognitive measures.

Exclusion Criteria:

1. Subjects with progressive MS.
2. Subjects with a contraindications for standard treatment with Rebif or Tecfidera including GI disease, needle phobia, liver disease.
3. Subjects treated with:

   * High dose intravenous immunoglobulin within 2 months prior to study entry
   * Natalizumab within 3 months prior to study entry
   * Immunosuppressive/immunomodulatory medications including cyclophosphamide, mitoxantrone, azathioprine, methotrexate, rituximab, ofatumumab, ocrelizumab, or alemtuzumab at any time.
4. Subjects with absolute lymphocyte count < 800 cells (mm3).
5. Subjects with any of the following neurologic/psychiatric disorder:

   * Severe depression during the past 12 months before screening;
   * History of substance abuse (treatment or alcohol) or any other factor (i.e., serious psychiatric condition) that may interfere with the subject's ability to cooperate and comply with the study procedures;
6. Subjects unable to undergo MRI scans, including claustrophobia or history of hypersensitivity to gadolinium-DTPA.
7. Pregnant or nursing females, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive HCG laboratory test.
8. Female subjects of childbearing potential, defined as all females physiologically capable of becoming pregnant, unless they agree to abstinence or, if sexually active, the use of contraception.
9. History of hypersensitivity to any of the study treatments or to treatments of similar chemical classes.
10. Subjects with abnormal Liver Function Test (LFT) levels

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a single center study conducted at the Partners Multiple Sclerosis Center. Patients who are planning to start a new disease modifying treatment for relapsing-remitting MS will be offered enrollment in this study of two commonly used MS treatments by their treating physician. Potential subjects will undergo inclusion/exclusion review by the study nurse. Those meeting criteria will be enrolled by overall study PI or treating physician. Subjects will be identified from the Partners MS Center at the Brigham and Women's Hospital. Potential subjects will initially be approached by their treating physician concerning the study.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-05; Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
T2 lesion load: Rebif v. Tecfidera | 6 months
  To compare two commonly used MS medications, IFN β-1a subcutaneous three times per week (Rebif) and oral twice daily dimethyl fumarate (Tecfidera), on mean number of new or enlarging T2 lesions at 6 months in adults with relapsing-remitting multiple sclerosis who are prescribed these medications and receive a 6 month MRI scan as standard of care.

SECONDARY OUTCOMES:
Reducing lesion load and MRI characteristics: Rebif v. Tecfidera | 6 months
  To compare Rebif vs. Tecfidera in reducing the T2 lesion volume, number of T1 black holes, gadolinium-enhancing lesions, brain parenchymal fraction, brain white matter fraction and brain gray matter fraction on the 6 month MRI.

CONTACTS AND LOCATIONS:
Locations (1):
- Partners MS Center, 1 Brookline Place Suite 225, Brookline, Massachusetts, United States

REFERENCES:
- [Background] Klawiter EC, Cross AH, Naismith RT. The present efficacy of multiple sclerosis therapeutics: Is the new 66% just the old 33%? Neurology. 2009 Sep 22;73(12):984-90. doi: 10.1212/WNL.0b013e3181b9c8f7. PMID 19770475
- [Background] Freedman MS, Hughes B, Mikol DD, Bennett R, Cuffel B, Divan V, LaVallee N, Al-Sabbagh A. Efficacy of disease-modifying therapies in relapsing remitting multiple sclerosis: a systematic comparison. Eur Neurol. 2008;60(1):1-11. doi: 10.1159/000127972. Epub 2008 Apr 25. PMID 18437041
- [Background] Randomised double-blind placebo-controlled study of interferon beta-1a in relapsing/remitting multiple sclerosis. PRISMS (Prevention of Relapses and Disability by Interferon beta-1a Subcutaneously in Multiple Sclerosis) Study Group. Lancet. 1998 Nov 7;352(9139):1498-504. PMID 9820297
- [Background] Kappos L, Gold R, Miller DH, Macmanus DG, Havrdova E, Limmroth V, Polman CH, Schmierer K, Yousry TA, Yang M, Eraksoy M, Meluzinova E, Rektor I, Dawson KT, Sandrock AW, O'Neill GN; BG-12 Phase IIb Study Investigators. Efficacy and safety of oral fumarate in patients with relapsing-remitting multiple sclerosis: a multicentre, randomised, double-blind, placebo-controlled phase IIb study. Lancet. 2008 Oct 25;372(9648):1463-72. doi: 10.1016/S0140-6736(08)61619-0. PMID 18970976
- [Background] Fox RJ, Miller DH, Phillips JT, Hutchinson M, Havrdova E, Kita M, Yang M, Raghupathi K, Novas M, Sweetser MT, Viglietta V, Dawson KT; CONFIRM Study Investigators. Placebo-controlled phase 3 study of oral BG-12 or glatiramer in multiple sclerosis. N Engl J Med. 2012 Sep 20;367(12):1087-97. doi: 10.1056/NEJMoa1206328. PMID 22992072
- [Background] Gold R, Giovannoni G, Phillips JT, Fox RJ, Zhang A, Meltzer L, Kurukulasuriya NC. Efficacy and safety of delayed-release dimethyl fumarate in patients newly diagnosed with relapsing-remitting multiple sclerosis (RRMS). Mult Scler. 2015 Jan;21(1):57-66. doi: 10.1177/1352458514537013. Epub 2014 Jul 2. PMID 24990854
- [Background] Gold R, Kappos L, Arnold DL, Bar-Or A, Giovannoni G, Selmaj K, Tornatore C, Sweetser MT, Yang M, Sheikh SI, Dawson KT; DEFINE Study Investigators. Placebo-controlled phase 3 study of oral BG-12 for relapsing multiple sclerosis. N Engl J Med. 2012 Sep 20;367(12):1098-107. doi: 10.1056/NEJMoa1114287. PMID 22992073
- [Background] Rudick RA, Lee JC, Simon J, Ransohoff RM, Fisher E. Defining interferon beta response status in multiple sclerosis patients. Ann Neurol. 2004 Oct;56(4):548-55. doi: 10.1002/ana.20224. PMID 15389896
- [Background] Wei X, Warfield SK, Zou KH, Wu Y, Li X, Guimond A, Mugler JP 3rd, Benson RR, Wolfson L, Weiner HL, Guttmann CR. Quantitative analysis of MRI signal abnormalities of brain white matter with high reproducibility and accuracy. J Magn Reson Imaging. 2002 Feb;15(2):203-9. doi: 10.1002/jmri.10053. PMID 11836778
- [Background] Liu L, Meier D, Polgar-Turcsanyi M, Karkocha P, Bakshi R, Guttmann CR. Multiple sclerosis medical image analysis and information management. J Neuroimaging. 2005;15(4 Suppl):103S-117S. doi: 10.1177/1051228405282864. PMID 16385023